CLINICAL TRIAL: NCT01509040
Title: Washington Study of Hemofiltration After Out-of-Hospital Cardiac Arrest
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Graham Nichol, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WASH CARDIAC
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Cardiac Arrest
Keywords: Resuscitated from Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Initiate standard post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Interventions: Other: Standard Care
- Low Volume Hemofiltration (Experimental): Initiate standard post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 45 mL/kg/h. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Interventions: Other: Standard Care; Device: Low Volume Hemofiltration
- High Volume Hemofiltration (Experimental): Initiate standard post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/kg/h, ultrafiltration 90 mL/kg/h. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Interventions: Other: Standard Care; Device: High Volume Hemofiltration

INTERVENTIONS:
Other: Standard Care — Triple-lumen central venous catheter inserted for pressure monitoring. All patients to receive 500-mL bolus of intravenous crystalloid every 30 minutes to achieve central venous pressure of 8 to 12 mm Hg; vasopressors if mean arterial pressure less than 65 mm Hg; and vasodilators if mean arterial pressure is 90 mm Hg or above.
  Initiation and maintenance of therapeutic hypothermia, target core temperature of below 34°C via standard external cooling techniques.
  Percutaneous coronary intervention performed as soon as feasible in patients with ST elevation or left bundle branch block on initial ECG.
  Serum biochemistry (including sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate) monitored every 6 hours.
Device: Low Volume Hemofiltration — Patients will receive isovolemic HF at a blood flow rate of 250 mL/min and ultrafiltration rate of 45 mL/kg/h for 48 hours. Initial replacement solution will be Prismasol BGK4/2.5. 3.1mg/dL phosphate (1.0 mmol/L) added to each bag. Replacement fluid adjusted as required based on chemistry values for sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution used. HF 1400 (i.e. polysulfone -based membrane) filters used throughout study. Hemofilter changed every 6 h after initiation of HF, and as required.
  Arms: Low Volume Hemofiltration
Device: High Volume Hemofiltration — Patients allocated to high volume HF will receive HF at 250 mL/h blood flow rate and 90 mL/kg/h ultrafiltration rate for 48 hours. All other care will be identical to that provided in the low volume HF group.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused into the bloodstream before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution will be used. HF 1400 (i.e. polysulfone -based membrane) filters will be used throughout the study. The hemofilter will be changed every 6 h after initiation of HF, and otherwise as required.
  Arms: High Volume Hemofiltration

SUMMARY:
The purpose of this study is to assess the feasibility of hemofiltration in patients resuscitated from cardiac arrest. Cardiac arrest is the loss of mechanical activity of the heart including the loss of detectable pulse, or spontaneous breathing. When heart function is restored, the cells of the body release molecules into the blood that cause inflammation, unstable blood pressure, organ dysfunction and death. Hemofiltration is a technique of washing the blood to remove fluid and molecules from it. Hemofiltration is a proven therapy for renal failure, but is considered investigational for treatment after resuscitation from cardiac arrest. Some experts believe that hemofiltration after heart function is restored can remove inflammation from the blood, maintain blood pressure and organ function. Others believe that intravenous fluid and medications are sufficient to maintain blood pressure and organ function. Since the inflammation that occurs after restoration of heart function lasts, the investigators continue hemofiltration for up to 48 hours. Whether hemofiltration or intravenous fluids and medications is better is not known. The investigators are checking if they can wash the blood of patients resuscitated from cardiac arrest before the investigators can begin a large randomized trial to test whether hemofiltration improves their outcome.

The investigators are testing this by randomly allocating patients resuscitated from cardiac arrest to receive low volume hemofiltration, high volume hemofiltration, or intravenous fluids and medications alone. The null hypotheses are that less than 80% of eligible patients will be enrolled, and that less than 80% of enrolled patients will undergo low-volume or high-volume hemofiltration (HF) for at least 80% of 48 hours.

DETAILED DESCRIPTION:
Patients resuscitated from out-of-hospital cardiac arrest will be randomly allocated to one of three groups; Standard of care: Initiate standard of post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Fluids, inotropes, vasopressors, vasodilators to maintain hemodynamics.

Low-volume Hemofiltration for 48 hours: Initiate standard of post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via a 11.5F double lumen venous catheter, blood flow 250mL/h, ultrafiltration 45mL/kg/h. Fluids, inotropes, vasopressors, vasodilators to maintain hemodynamics.

High-volume Hemofiltration for 48 hours: Initiate standard of post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 90 mL/kg/h. Fluids, inotropes, vasopressors, vasodilators to maintain hemodynamics.

30 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* adults
* restoration of spontaneous circulation sustained to hospital arrival after OOHCA with any first recorded rhythm
* aged >=65 years
* less than 1 h from call to 911 until emergency department arrival
* less than 6 h from arrival until randomization
* informed consent provided by legally-authorized representative

Exclusion Criteria:

* do not attempt resuscitation orders; known end-stage terminal illness pre-arrest; major pre-arrest neurological dysfunction; another reason to be comatose (e.g. drug overdose)
* chronic steroid use
* non-English speaking LAR
* previous enrollment in the trial
* blunt, penetrating, or burn-related injury; exsanguination; drowning, electrocution or strangulation
* known pregnancy
* known prisoner
* weight > 100 kg
* persistent (i.e. 30 minutes) SBP< 80 mmHg despite pressors; refractory ventricular arrhythmias; severe bradycardia without a pacemaker
* thrombocytopenia (i.e. < 50,000/microL) or coagulopathy (i.e. INR > 1.5) or inferior vena cava filter in situ
* known cirrhosis
* serum ionized calcium < 2.2 mmol/L serum lactate > 6 mmol/L
* obeying verbal commands

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Nichol, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control group: Initiate standard post-resuscitative care including triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious via standard external cooling techniques. Fluids, 500-mL bolus of intravenous crystalloid every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Percutaneous coronary intervention performed as soon as feasible in patients with ST elevation or left bundle branch block on initial ECG.
  Serum biochemistry (including sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate) monitored every 6 hours.
- Low Volume Hemofiltration: Low Volume Hemofiltration: Initiate standard post-resuscitative care as in control group. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 45 mL/kg/h.
  Low Volume Hemofiltration: Patients will receive isovolemic HF. Initial replacement solution will be Prismasol BGK4/2.5. 3.1mg/dL phosphate (1.0 mmol/L) added to each bag. Replacement fluid adjusted as required based on chemistry values for sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution used. HF 1400 (i.e. polysulfone -based membrane) filters used throughout study. Hemofilter changed every 6 h after initiation of HF, and as required.
- High Volume Hemofiltration: High Volume Hemofiltration: Initiate standard post-resuscitative care as in control group. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/kg/h, ultrafiltration 90 mL/kg/h. .
  High Volume Hemofiltration: Patients allocated to high volume HF will receive HF at 250 mL/h blood flow rate and 90 mL/kg/h ultrafiltration rate for 48 hours. All other care will be identical to that provided in the low volume HF group.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused into the bloodstream before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution will be used. HF 1400 (i.e. polysulfone -based membrane) filters will be used throughout the study. The hemofilter will be changed every 6 h after initiation of HF, and otherwise as required.
Period: Overall Study
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Started | 0 | 2 | 0
Completed | 0 | 1 | 0
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration | Total
Number analyzed (Participants) | 0 | 2 | 0 | 2
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 |  | 0
  Between 18 and 65 years |  | 0 |  | 0
  >=65 years |  | 2 |  | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] |  | 67 [65 to 69] |  | 67 [65 to 69]
Gender [Number; unit: participants]
  Female |  | 1 |  | 1
  Male |  | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Intervention Compliance
Description: Intervention Compliance will be defined as the proportion of intervention patients who are alive and undergo hemofiltration (HF) for at least 80% of 48 hours from randomization.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 1 |

2. Secondary Outcome: Enrollment
Description: This will be defined as the proportion of eligible patients who are randomized.
Time Frame: 12 hours
Measure: Number; unit: participants
Groups:
- Control: Initiate standard post-resuscitative care including triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Standard Care: Triple-lumen central venous catheter inserted for pressure monitoring. All patients to receive 500-mL bolus of intravenous crystalloid every 30 minutes to achieve central venous pressure of 8 to 12 mm Hg; vasopressors if mean arterial pressure less than 65 mm Hg; and vasodilators if mean arterial pressure is 90 mm Hg or above.
  Initiation and maintenance of therapeutic hypothermia, target core temperature of below 34°C via standard external cooling techniques.
  Percutaneous coronary intervention performed as
- Low Volume Hemofiltration: Initiate standard post-resuscitative care including triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 45 mL/kg/h. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Standard Care: Triple-lumen central venous catheter inserted for pressure monitoring. All patients to receive 500-mL bolus of intravenous crystalloid every 30 minutes to achieve central venous pressure of 8 to 12 mm Hg; vasopressors if mean arterial pressure less than 65 mm Hg; and vasodilators if mean arterial pressure is 90 mm Hg or above.
  Initiation and maintenance of therapeutic hypothermia, target core tem
- High Volume Hemofiltration: Initiate standard post-resuscitative care including a triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/kg/h, ultrafiltration 90 mL/kg/h. Fluids, 500-mL bolus of intravenous crystalloid given every 30 minutes to achieve a central venous pressure of 8 to 12 mm Hg; inotropes, vasopressors if mean arterial pressure is less than 65 mm Hg; vasodilators, if mean arterial pressure is 90 mm Hg or above to maintain hemodynamics.
  Standard Care: Triple-lumen central venous catheter inserted for pressure monitoring. All patients to receive 500-mL bolus of intravenous crystalloid every 30 minutes to achieve central venous pressure of 8 to 12 mm Hg; vasopressors if mean arterial pressure less than 65 mm Hg; and vasodilators if mean arterial pressure is 90 mm Hg or above.
  Initiation and maintenance of therapeutic hypothermia, target core
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 2 |

3. Secondary Outcome: Clearance of Inflammatory Mediators
Description: Venous blood samples will be obtained periodically after randomization, processed, stored, then tested for serum cytokine levels.
Time Frame: 48 hours
Population: The outcome was not assessed.
Groups:
- Control: Control group: Initiate standard post-resuscitative care including triple lumen catheter to monitor central venous pressure, core temperature maintenance between 32C and 34C if unconscious via standard external cooling techniques. Fluids, 500-mL bolus of intravenous crystalloid every 30 minutes to achieve a central venous pressure of 8 to 12 mmHg; inotropes, vasopressors if mean arterial pressure is less than 65 mmHg; vasodilators, if mean arterial pressure is 90 mmHg or above to maintain hemodynamics.
  Percutaneous coronary intervention performed as soon as feasible in patients with ST elevation or left bundle branch block on initial ECG.
  Serum biochemistry (including sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate) monitored every 6 hours.
- Low Volume Hemofiltration: Low Volume Hemofiltration: Initiate standard post-resuscitative care as in control group. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 45 mL/kg/h.
  Low Volume Hemofiltration: Patients will receive isovolemic HF. Initial replacement solution will be Prismasol BGK 4/2.5. 3.1mg/dL phosphate (1.0 mmol/L) added to each bag. Replacement fluid adjusted as required based on chemistry values for sodium, potassium, bicarbonate, glucose, calcium, phosphate, magnesium and lactate.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution used. HF 1400 (i.e. polysulfone-based membrane) filters used throughout study. Hemofilter changed every 6h after initiation of HF, and as required.
- High Volume Hemofiltration: High Volume Hemofiltration: Initiate standard post-resuscitative care as in control group. Hemofiltration x 48 hours via 11.5F double lumen venous catheter, blood flow 250 mL/h, ultrafiltration 90 mL/kg/h.
  HIgh Volume Hemofiltration: Patients allocated to high volume HF will receive HF at 250 mL/h blood flow rate and 90 mL/kg/h ultrafiltration rate for 48 hours. All other care will be identical to that provided in the low volume HF group.
  Vascular access for HF will be via an 11.5-F, double-lumen venous catheter in a central vein. The hemofiltrate will be replaced by fluid infused into the bloodstream before (i.e. predilution) and after (i.e. postdilution) the filter. A fixed ratio of 80:20 predilution:postdilution will be used. HF 1400 (i.e. polysulfone-based membrane) filters used throughout study. Hemofilter changed every 6h after initiation of HF, and as required.
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Total Volume Intravenous Fluid Infused
Description: This will be defined as the volume of fluid (in mL) infused during the first 48 hours from enrollment.
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: mL
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
mL |  | 10652.5 [8043 to 13262] |

5. Secondary Outcome: Use of Pressors and Inotropes
Description: This includes use of dopamine, dobutamine, epinephrine, nesiritide, norepinephrine, or phenylephrine during the first 48 hours from enrollment.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 1 |

6. Secondary Outcome: Shock
Description: This will be defined as systolic blood pressure < 65 at the end of any four hour period during the initial 48 hours of enrollment in control and intervention patients.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 0 |

7. Secondary Outcome: Ejection Fraction
Description: This will be assessed by standard transthoracic echocardiographic methods 48 hours after enrollment in control and intervention patients
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: percentage
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
percentage |  | 65 [55 to 75] |

8. Secondary Outcome: Number of Hospital Days
Description: This will be described for all hospitalized patients as a measure of morbidity after resuscitation.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
days |  | 8.5 [2 to 15] |

9. Secondary Outcome: Time Interval From 911 Call to Patient Death
Description: This will be described for all hospitalized patients as a measure of morbidity after resuscitation.
Time Frame: 1 year
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
Days |  | 183.6 [2.2 to 365] |

10. Secondary Outcome: Expected Adverse Event
Description: Device-Related Hematoma at insertion site, vessel perforation, wound infection, deep venous thrombosis or pulmonary embolism.
  Device Failure Mechanical failure Hypertension- SBP>160 mmHg, or DBP >120 mmHg. Hypotension- SBP<60 mmHg. Hypervolemia- CVP > 12 cm. Hypovolemia- CVP < 2 cm. Hypokalemia- serum potassium concentration < 3.5 mmol/L. Alkalosis- serum bicarbonate > 32 mmol/L. Hyperglycemia- serum glucose > 240 mg/dL. Hypophosphatemia- serum phosphate concentration < 0.8 mmol/L. Hypocalcemia- serum ionized calcium < 2.2 mmol/L. Lactic acidosis- serum lactate > 6 mmol/L.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 2 |

11. Secondary Outcome: Safety Outcome, Number of Participants With STEMI, Radiographic Pulmonary Edema, or Arrhythmia
Description: ST-Elevation Myocardial Infarction- ECG criteria and biomarker criteria for acute infarction.
  Radiographic Pulmonary Edema- radiographic presence of alveolar or interstitial edema, bilateral pleural effusions, cardiomegaly or venous congestion.
  Arrhythmia- other than sinus rhythm observed after randomization. Arrhythmia requiring treatment- rhythm with subsequent use of an antiarrhythmic drug or electrical therapy observed after randomization.
  Arrhythmia with cardiovascular instability- any rhythm with cardiovascular instability as determined by the DSMB, observed after randomization.
Time Frame: 48 hours
Measure: Number; unit: Participant
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
Participant |  | 2 |

12. Secondary Outcome: Unexpected Adverse Device Events (UADE)
Description: These will be defined as any unexpected adverse effect on health or safety or any unexpected life-threatening problem caused by, or associated with, a device, if that effect or problem was not previously identified in nature, severity, or degree of incidence in this investigation plan or application which will be submitted to the Food and Drug Administration (including a supplementary plan or application), or any other unexpected serious problem associated with a device. The death or neurological impairment of an individual patient will not be considered an adverse event in this study.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 0 |

13. Secondary Outcome: Clinical Safety Outcomes; Number of Participants With Clinical Diagnoses
Description: Clinical diagnoses of cerebral bleeding, stroke, bleeding requiring transfusion or surgical intervention, rearrest, pulmonary edema, rib or sternal fractures, internal thoracic or abdominal injuries as noted in the discharge summary
Time Frame: Discharge
Measure: Number; unit: participants
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Number analyzed (Participants) | 0 | 2 | 0
participants |  | 2 |

ADVERSE EVENTS:
Arm/Group | Control | Low Volume Hemofiltration | High Volume Hemofiltration
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=0) | Low Volume Hemofiltration (N=2) | High Volume Hemofiltration (N=0)
Arrhythmia associated with cardiovascular instability (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=0) | Low Volume Hemofiltration (N=2) | High Volume Hemofiltration (N=0)
Arrhythmia associated with low blood pressure (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes